CLINICAL TRIAL: NCT05015517
Title: Comparison of Ultrasound Guided Erector Spinae Block and Supra-inguinal Fascia Iliaca Block for Postoperative Analgesia in Patients Undergoing Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: ESP Block vs FIB in Patients Undergoing Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abdallah Moawad, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ESP vs FIB in hip arthroplasty
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hip Arthropathy
Keywords: Erector spinae block; Fascia iliaca block

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: computer-generated sequence. Concealment will be achieved using opaque envelopes. All data will be collected blindly and the authors will perform the blocks without interference in data collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB Group (Active Comparator): This group will receive ultrasound-guided erector spinae plane block and subarachnoid block.
  Interventions: Procedure: Erector spinae plain block
- FIB Group (Active Comparator): This group will receive supra-inguinal fascia iliaca block and subarachnoid block .
  Interventions: Procedure: Fascia Iliaca block

INTERVENTIONS:
Procedure: Erector spinae plain block — Patients will be placed in the lateral position.Ultrasonography will be performed by an experienced anesthetist.The 4th lumbar vertebral level will be determined using the conventional method (imaginary line between two iliac crests). The low frequency convex probe (2-5MHz) will then be placed at the mid-vertebral line in the sagittal plane. It will be shifted from the midline, 3.5-4 cm lateral to the side of the surgery to visualize the erector spinae muscle and transverse process. Using the out-plane technique a 22G/80-mm block needle will be advanced until it reaches the transverse process. After negative aspiration, 0.5-1 ml of the prepared local anaesthetic solution (20 ml bupivacaine 0.5%, 10 ml lidocaine 2%) and 10 ml normal saline will be administered for hydrodissection to confirm correct location. The needle will be repositioned by pulling back a few millimeters if resistance occurred when injecting local anesthesia
  Arms: ESPB Group
Procedure: Fascia Iliaca block — Patients will be placed in supine position. Ultrasonography will be performed by an experienced anesthetist using ultrasound device equipped with a low frequency (2-5 MHz) convex probe and an echogenic 21 G/ 10 cm needle will be used.
  The probe will be placed in the inguinal crease. Scan will be started laterally from the femoral artery and nerve in the inguinal crease to identify the Sartorius muscle. The muscle will then be traced until its origin at the anterior superior iliac spine is identified and the shadow of the bony of iliac crest & iliacus muscle will be seen. Injection will be performed at the plane deep to the fascia iliaca and above the lateral part of the iliacus muscle. After negative aspiration, the prepared local anaesthetic solution (15 ml bupivacaine 0.5%, 15 ml normal saline) will be injected incrementally, aspirating every 5 ml.
  Arms: FIB Group

SUMMARY:
The aim of this study is to compare between the analgesic efficacy of ESP block and FIB in patients undergoing hip arthroplasty.

DETAILED DESCRIPTION:
Hip arthroplasty surgery is usually associated with severe postoperative pain. Several modalities are usually used for postoperative analgesia in these patients, those include; intravenous analgesia, neuraxial analgesia and peripheral nerve blocks.

Peripheral nerve blocks have several advantages such as; potent analgesia, lower motor impairment and minimal systemic complications.

Lumbar plexus block and supra-inguinal fascia iliaca block (FIB) are the most commonly performed peripheral nerve blocks for hip surgeries.

Fascia iliaca block is one of the most common techniques for pain control after hip surgeries; it can be regarded as an anterior approach of the lumbar plexus. It provides analgesia through spread of local anaesthetic to the femoral and lateral cutaneous femoral nerves.

Ultrasound guided erector spinae plane (ESP) block is a recent regional anesthetic technique. It was first described in 2016 for acute and chronic thoracic pain management. It is a paraspinal fascial plane block that provides analgesia through injecting local anesthetic drugs to block the ventral and dorsal rami of spinal nerves in the paravertebral area.

To the best of the investigators knowledge, the use of ESP block in hip surgery was only investigated in one study and few case reports. Therefore, further randomized controlled studies are needed to prove this hypothesis.

This study aims to investigate the efficacy of ESP block in hip replacement compared to the supra-inguinal FIB.

The investigators hypothesize that erector spinae block may provide better postoperative analgesia than fascia iliaca block, since erector spinae block provides analgesic cover for the entire lumbar plexus rather than just peripheral nerves provided by fasicia iliaca.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* ASA grade I to II
* Patients scheduled for hip replacement surgeries under subarachnoid block (SAB) e.g. hip hemi-arthroplasty, total hip arthroplasty

Exclusion Criteria:

* Patient refusal
* Age below 18 or above 65 years.
* ASA grade III to IV
* Patients with known allergies to any of the drugs used.
* Contraindication to SAB eg. Coagulopathy, infection at the injection site, severe cardiopulmonary disease, diabetic or other neuropathies.
* Patients receiving opioids for chronic analgesic therapy
* Inability to comprehend visual analogue scale (VAS)
* Infection at site of erector spinae or fascia iliaca block.
* Body mass index >35 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Total morphine requirements | 24 hours postoperatively
  Amount of morphine required postoperatively

SECONDARY OUTCOMES:
Visual analogue pain score | at rest at 2, 4, 6, 12, 18, and 24 hours postoperatively
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Time to first postoperative analgesic request | 24 hours postoperatively
  If the visual analogue scale (VAS) was 4 or more, a morphine increment (2 mg) will be added to maintain a resting VAS at <3 and the total 24-hours morphine consumption will be recorded.
Quadriceps muscle power strength | at 6, 12 and 24 hours postoperatively
  For motor block assessment, the patient knee will be fully flexed and the patient will be asked to extend it. The motor block will be classified as follows: grade 0; normal muscle power, grade 1; motor weakness, grade 2; complete motor paralysis

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf RA Aswa, Professor, Study Director — Cairo University

REFERENCES:
- See also: Continuous psoas compartment block for postoperative analgesia after total hip arthroplasty: new landmarks, technical guidelines, and clinical evaluation — https://journals.lww.com/anesthesia-analgesia/fulltext/2002/06000/continuous_psoas_compartment_block_for.45.aspx
- See also: Abrahams MS, Aziz MF. Ambulatory continuous posterior lumbar plexus blocks following hip arthroscopy: a review of 213 cases — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=+Nye+ZB%2C+Horn+JL%2C+Crittenden+W%2C+Abrahams+MS%2C+Aziz+MF.+Ambulatory+continuous+posterior+lumbar+plexus+blocks+following+hip+arthroscopy%3A+a+review+of+213+cases.%C2%A0J+Clin+Anesth.%C2%A02013+Jun%3B25%284%29%3A268-274.++Bullock+WM&btnG=#d=gs_qabs&u=%23p%3DCrp2CiuaHgMJ
- See also: Ultrasound-Guided Suprainguinal Fascia Iliaca Technique Provides Benefit as an Analgesic Adjunct for Patients Undergoing Total Hip Arthroplasty — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Bullock+WM%2C%C2%A0Yalamuri+SM%2C%C2%A0Gregory+SH%2C%C2%A0Auyong+DB%2C%C2%A0Grant+SA%2C+Ultrasound-Guided+Suprainguinal+Fascia+Iliaca+Technique+Provides+Benefit+as+an+Analgesic+Adjunct+for+Patients+Undergoing+Total%C2%A0Hip%C2%A0Arthroplasty%2C+J+Ultrasound+Med.%2C+2017+Feb%3B36%282%29%3A433-438.&btnG=#d=gs_qabs&u=%23p%3DNHm8V774Mx0J
- See also: Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=Desmet%C2%A0M%2C%C2%A0Vermeylen%C2%A0K%2C%C2%A0Van+Herreweghe%C2%A0I%2C+et+al.A+Longitudinal+Supra-Inguinal+Fascia+Iliaca+Compartment+Block+Reduces+Morphine+Consumption+After+Total+Hip+Arthroplasty.Regional+Anesthesia+%26Pain+Medicine%C2%A02017%3B42%3A327-333.&btnG=#d=gs_qabs&u=%23p%3D4cdBlf-qnskJ
- See also: The erector spinae plane block: a novel analgesic technique in thoracic neuropathic pain. — https://scholar.google.com/scholar?hl=en&as_sdt=0%2C5&q=++Forero+M%2C+Adhikary+SD%2C+Lopez+H%2C+et+al.+The+erector+spinae+plane+block%3A+a+novel+analgesic+technique+in+thoracic+neuropathic+pain.+Reg+Anesth+Pain+Med.+2016%3B41%285%29%3A621%E2%80%93627.&btnG=#d=gs_qabs&u=%23p%3DFSUO-gw42YEJ
- See also: Erector spinae plane block an effective block for postoperative analgesia in modified radical mastectomy. — https://search.proquest.com/openview/70d234ac1634867694810005281fe12a/1?pq-origsite=gscholar&cbl=226517